CLINICAL TRIAL: NCT02553876
Title: An Observational Cohort Study to Assess the Long Term Effectiveness of Dorsal Root Ganglion Stimulation for Chronic Pain in the Upper Limb(s)
Brief Title: Dorsal Root Ganglion Stimulation for Hand and Upper Limb Pain
Status: Terminated | Type: Observational
Why Stopped: Stopped 1 jan 2017, logistical reasons
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Diakonessenhuis, Utrecht (Other)
Responsible Party: Principal Investigator, Jennifer Breel, Research coordinator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: AMS-01-2015
Record Dates: First submitted 2015-09-02; First posted 2015-09-18 (Estimated); Last update posted 2021-12-14 (Actual); Status verified 2021-11

CONDITIONS: Dorsal Root Ganglion Stimulation; Pain in Limb, Hand, Foot, Fingers and Toes; Causalgia of Upper Limb
Keywords: neurostimulation; dorsal root ganglion; hand pain; upper limb pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational: All patients referred with pain in the hand and/or upper limb will be evaluated. Patients will first be assessed for suitability for neurostimulation implantation and then included in the study. Patients wiil fill in questionnaires (pain scores, Quality of Life and satisfaction) at baseline and post-operatively at regular intervals (as per standard of care in the Netherlands.)

SUMMARY:
There are no studies as yet specifically investigating the application of DRG stimulation in the treatment of chronic pain affecting the upper limbs. The investigators propose to investigate the effect of dorsal root stimulation in patients with chronic hand or upper limb pain.

DETAILED DESCRIPTION:
Dorsal Root Ganglion (DRG) stimulation is a form of Spinal Cord Stimulation (SCS), which has been available and used for the treatment of chronic pain in Europe since late 2011. Clinical practice and pre/post market studies have shown that stimulation of the DRG can significantly reduce chronic intractable pain of various aetiologies. However, there are no studies as yet specifically investigating the application of DRG stimulation in the treatment of chronic pain affecting the upper limbs. Furthermore, there are very few studies of SCS generally, in an upper limb pain population, despite this being a group often referred for and treated with SCS in tertiary, interventional pain practices. Due to several limitations of traditional SCS systems, chiefly concerning the stability of stimulation induced paraesthesia, DRG stimulation is being increasingly utilised in its place for this condition.

ELIGIBILITY:
* Subject is appropriate for SCS implantation according to standard criteria from the Dutch Neuromodulation Society
* Subject is >18 to <75 years old.
* Subject is able and willing to comply with the follow-up schedule and protocol
* Subject has chronic (> 6 months) uni/bi-lateral pain, primarily in the upper limb(s)
* (Arm and/or Hand)
* Minimum baseline pain rating of 60 mm on the VAS in the primary region of pain
* Documented, successful paraesthesia mapping of transient stimulation over painful anatomy
* Subject is able to provide written informed consent

Exclusion criteria

* Subject has no other exclusion criteria for SCS implantation according to standard criteria from the Dutch Neuromodulation Society
* Subject has had corticosteroid therapy at an intended site of stimulation within the past 30 days
* Subject has had radiofrequency treatment of an intended target DRG within the past 3 months
* Subject has participated in another clinical study within 30 days
* Subject has been previously treated with and failed to respond to an implantable neuromodulation therapy
* Subject has had a complete or partial amputation of the painful upper limb(s) and is experiencing phantom and/or stump pain post amputation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Twenty (20) subjects of either gender, minimum of 18 years of age, maximum of 75 years of age, suffering from chronic, refractory upper limb pain for at least 6 months, who have been or will be routinely scheduled to receive the commercially available DRG Neurostimulator System.
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Pain reduction | 5 years
  Pain measured on a 10cm Visual Analogue Scale (VAS), where 0 [no pain] and 10 [worst possible pain] imaginable

SECONDARY OUTCOMES:
Comfort of stimulation | 5 years
  Via novel questionnaire patient will validate sensation of paresthesia in different body positions
Quality of life | 5 years
  EuroQol-5D, Short Form-36
Sleep Quality | 5 years
  Using novel Amsterdam Sleep Questionnaire for patients with a neurostimulator
Subject satisfaction | 5 years
  Global Perceived Effect Scale
Pain medication utilization | 5 years
  Medication usage before and after implantation will be registered
Safety | 5 years
  Long term follow up of device related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Markus W Hollmann, MD, PhD, Principal Investigator — Principal Investigator
Locations (3):
- Netherlands (3):
  - Noordwest Ziekenhuisgroep, Alkmaar, North Holland
  - Academic Medical Center, Amsterdam, North Holland
  - Diakonessenhuis, Zeist, Utrecht